CLINICAL TRIAL: NCT05610176
Title: BIO|CONCEPT.Amvia, First in Human Study for the Amvia/Solvia Pacemaker Family
Brief Title: BIO|CONCEPT.Amvia Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik Australia Pty Ltd. (Industry)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Organization: Biotronik SE & Co. KG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA115
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-06

CONDITIONS: Bradycardia; Heart Failure
Keywords: Cardiac pacemaker; CRT-P
MeSH Terms: conditions — Bradycardia; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amvia Sky pacemaker or CRT-P implantation (Experimental): Patients implanted with an Amvia Sky pacemaker or CRT-P device
  Interventions: Device: Amvia Sky pacemaker or CRT-P device

INTERVENTIONS:
Device: Amvia Sky pacemaker or CRT-P device — Subjects with an indication for a pacemaker or CRT-P device will be implanted with an Amvia Sky device of the Amvia/Solvia pacemaker family according to standard pacemaker implantation procedures. Device programming will be done according to the medical needs of the subjects.

SUMMARY:
The goal of this exploratory study is to test the preliminary safety and product performance of the new Amvia/Solvia pacemaker family in subjects that require a pacemaker or cardiac resynchronization therapy pacemaker (CRT-P) implantation. The study will be conducted at sites in Australia and New Zealand. It is planned to include 50 subjects in the study. Participants will visit sites at enrollment in the study, at implantation, pre-hospital discharge, 1- 3- and 12-month follow-up visits. At the visits the device will be interrogated and standard device measurements including those related to special features will be performed to assess the functionality of the device. Programming of the pacemakers will be done according to the participant´s therapeutical needs.

ELIGIBILITY:
Inclusion Criteria:

* Standard indication for pacemaker or cardiac resynchronization therapy pacemaker (CRT-P) implantation, including de novo, upgrade or replacement implantations
* Ability to understand the nature of the study
* Willingness to provide written informed consent
* Ability and willingness to perform all follow-up visits at the study site
* Ability and willingness to use the CardioMessenger and acceptance of the BIOTRONIK Home Monitoring concept

Exclusion Criteria:

* Planned for conduction system pacing
* Planned for activation of atrial anti-tachycardia pacing (aATP) without known history of atrial arrhythmia, or with permanent atrial fibrillation (AF)
* Planned cardiac surgical procedures or interventional measures other than the study procedure within the next 12 months
* Pregnant or breast feeding
* Age less than 18 years
* Participation in another interventional clinical investigation according to the definition given in the study protocol
* Life-expectancy less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Mariani, Dr, Principal Investigator — The Alfred
Locations (7):
- Australia (6):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Advara Heart Care Wesley, Auchenflower, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Peninsula Heart Centre, Frankston, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Christchurch Hospital, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 52 patients were enrolled between the date of first patient in (November 23, 2022) and last patient in (May 25, 2023).
  Patients that were already enrolled at the time of the notification of enrollment stop (after the 50th implantation) were still admitted for implantation, thus leading to two more patients than specified in the protocol (N=50)l.
Pre-assignment Details: 50 patients were planned to be enrolled according to the protocol. At the time of the notification of enrollment stop (after the 50th implantation), two additional patients were already enrolled, thus leading to a total of 52 enrolled patients.
  All enrolled patients provided written informed consent and were implanted with an investigational device.
Groups:
- Amvia Sky Pacemaker or CRT-P Implantation: Patients implanted with an Amvia Sky pacemaker or CRT-P device
  Amvia Sky pacemaker or CRT-P device: Subjects with an indication for a pacemaker or CRT-P device were implanted with an Amvia Sky device of the Amvia/Solvia pacemaker family according to standard pacemaker implantation procedures. After implantation with an investigational device, the patients were seen by the investigator at pre-hospital discharge, 1-month, 3-months, and 12-months follow-up. All clinical procedures were performed according to clinical routine.
Period: Overall Study
Arm/Group | Amvia Sky Pacemaker or CRT-P Implantation
Started | 52
Completed | 46
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | Amvia Sky Pacemaker or CRT-P Implantation
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasion | 49
  Ethnicity: Black | 0
  Ethnicity: Asian | 1
  Ethnicity: Indigenous | 1
  Ethnicity: Other | 1
Region of Enrollment [Number; unit: participants]
  Australia | 36
  New Zealand | 16

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Device Effect (SADE)-Free Rate After 12 Months
Description: Descriptive statistics of the investigational device related SADE-free rate after first implantation attempt will be calculated using a Kaplan-Meier estimate
Time Frame: 12 months
Population: All 52 patients implanted with an investigational device contribute to the analysis of the SADE-free rate.
  Neither any of the 46 patients with regular study termination after 12 months, nor any of the 6 patients with premature study termination had any SADE.
  Thus, a 95% CI for the SADE-free rate could methodologically not be estimated with the Kaplan-Meier method, but instead with the binomial method.
Measure: Count of Participants; unit: Participants
Arm/Group | Amvia Sky Pacemaker or CRT-P Implantation
Number analyzed (Participants) | 52
Participants | 52

2. Other Pre Specified Outcome: Right Atrial Sensing Amplitude
Description: The sensing amplitude is measured using a programmer device during the follow-up examination of a pacemaker patient. It refers to the minimum voltage of the heart's intrinsic electrical signals that a pacemaker can detect through its leads to monitor the heart's natural activity and decide whether pacing is needed. In this case refering to the lead placed in the right atrium.
Time Frame: 12 months
Population: The analysis population for right atrial lead parameters consists of those patients that were implanted with an atrial lead, i.e. patients with a dual- or triple-chamber device, and for whom a value was measured at the specified timepoint.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Amvia Sky Pacemaker or CRT-P Implantation
Number analyzed (Participants) | 39
mV | 3.4 (1.9)

3. Other Pre Specified Outcome: Right Atrial Pacing Threshold
Description: The pacing threshold is measured using a programmer device during the follow-up examination of a pacemaker patient. It refers to the minimum amount of electrical energy required to consistently depolarize the myocardium, thereby triggering a cardiac contraction. In this case refering to the lead placed in the right atrium.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: V
Arm/Group | Amvia Sky Pacemaker or CRT-P Implantation
Number analyzed (Participants) | 37
V | 0.9 (0.7)

4. Other Pre Specified Outcome: Right Ventricular Sensing Amplitude
Description: The sensing amplitude is measured using a programmer device during the follow-up examination of a pacemaker patient. It refers to the minimum voltage of the heart's intrinsic electrical signals that a pacemaker can detect through its leads to monitor the heart's natural activity and decide whether pacing is needed. In this case refering to the lead placed in the right ventricle.
Time Frame: 12 months
Population: The analysis population for right ventricular lead parameters consists of all patients for whom a value was measured at the specified timepoint.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Amvia Sky Pacemaker or CRT-P Implantation
Number analyzed (Participants) | 45
mV | 10.8 (3.9)

5. Other Pre Specified Outcome: Right Ventricular Pacing Threshold
Description: The pacing threshold is measured using a programmer device during the follow-up examination of a pacemaker patient. It refers to the minimum amount of electrical energy required to consistently depolarize the myocardium, thereby triggering a cardiac contraction. In this case refering to the lead placed in the right ventricle.
Time Frame: 12 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: V
Arm/Group | Amvia Sky Pacemaker or CRT-P Implantation
Number analyzed (Participants) | 46
V | 0.9 (0.3)

6. Other Pre Specified Outcome: Left Ventricular Sensing Amplitude
Description: The sensing amplitude is measured using a programmer device during the follow-up examination of a pacemaker patient. It refers to the minimum voltage of the heart's intrinsic electrical signals that a pacemaker can detect through its leads to monitor the heart's natural activity and decide whether pacing is needed. In this case refering to the lead placed next to the left ventricle.
Time Frame: 12 months
Population: The analysis population for left ventricular lead parameters consists of those patients that were implanted with an LV lead, i.e. patients with a triple-chamber device, and for whom a value was measured at the specified timepoint.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Amvia Sky Pacemaker or CRT-P Implantation
Number analyzed (Participants) | 7
mV | 11.5 (6.0)

7. Other Pre Specified Outcome: Left Ventricular Pacing Threshold
Description: The pacing threshold is measured using a programmer device during the follow-up examination of a pacemaker patient. It refers to the minimum amount of electrical energy required to consistently depolarize the myocardium, thereby triggering a cardiac contraction. In this case refering to the lead placed next to the left ventricle.
Time Frame: 12 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: V
Arm/Group | Amvia Sky Pacemaker or CRT-P Implantation
Number analyzed (Participants) | 7
V | 1.4 (0.5)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from enrollment until study exit at 12-month follow-up, i.e. for one year.
Arm/Group | Amvia Sky Pacemaker or CRT-P Implantation
All-Cause Mortality (participants affected / at risk) | 6/52
Serious Adverse Events (participants affected / at risk) | 30/52
Other Adverse Events (participants affected / at risk) | 27/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amvia Sky Pacemaker or CRT-P Implantation (N=52)
Pneumonia (Infections and infestations) | 4 (6)
Adverse drug reaction (General disorders) | 4 (5)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 3 (3)
Respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Delirium (Psychiatric disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (2)
Accelerated idioventricular rhythm (Cardiac disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Candida infection (Infections and infestations) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Condition aggravated (General disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Gastrooesophageal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Herpes simplex encephalitis (Infections and infestations) | 1 (1)
Herpes simplex meningoencephalitis (Infections and infestations) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Iliac artery perforation (Vascular disorders) | 1 (1)
Implant site erythema (General disorders) | 1 (1)
Implant site pain (General disorders) | 1 (1)
Implant site swelling (General disorders) | 1 (1)
Implant site warmth (General disorders) | 1 (1)
Inflammatory marker increased (Investigations) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Intestinal mass (Gastrointestinal disorders) | 1 (1)
Lead dislodgement (Product Issues) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Morganella infection (Infections and infestations) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia moraxella (Infections and infestations) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amvia Sky Pacemaker or CRT-P Implantation (N=52)
Device computer issue (Product Issues) | 5 (8)
Adverse drug reaction (General disorders) | 3 (4)
Corona virus infection (Infections and infestations) | 3 (3)
Angina pectoris (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 2 (2)
Device stimulation issue (Product Issues) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Gout (Metabolism and nutrition disorders) | 1 (2)
Left ventricular dysfunction (Cardiac disorders) | 1 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1)
Cardiac sarcoidosis (Cardiac disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Device programming error (Injury, poisoning and procedural complications) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gastrointestinal stoma output abnormal (Investigations) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Implant site haematoma (General disorders) | 1 (1)
Implant site pain (General disorders) | 1 (1)
Implant site paraesthesia (General disorders) | 1 (1)
Implant site swelling (General disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin candida (Infections and infestations) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1)
Undersensing (Product Issues) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (4):
  • Study Protocol: sections 1-9 (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT05610176/Prot_000.pdf
  • Study Protocol: sections 10-23 (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT05610176/Prot_001.pdf
  • Study Protocol: Amendments (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT05610176/Prot_002.pdf
  • Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT05610176/SAP_003.pdf